CLINICAL TRIAL: NCT06812572
Title: A Prospective Clinical Study to Evaluate the Repeatability of the Visibly Vision Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visibly (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VVT-1002
Record Dates: First submitted 2019-03-05; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: multi-center, single-arm, non-randomized, non-blinded, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1 (Other): Without using an available refractive correction and whose refractive error is no greater than -1.00D of myopia (spherical component in minus cylinder format) and with no greater than -2.00D of astigmatism in either eye
  Interventions: Device: Visibly Vision Test
- Cohort 2 (Other): With prior correction of no greater than -6.00D of myopia (spherical component in minus cylinder format) and require a spherical (non-astigmatic) over-refraction of no more than ±1.00 D in either eye
  Interventions: Device: Visibly Vision Test

INTERVENTIONS:
Device: Visibly Vision Test — The Visibly Vision Test is used as a digital self-administered device to measure visual acuity and to subjectively measure refractive value for a patient's eye to determine the optical prescription for the conditions of myopia and astigmatism

SUMMARY:
The study is a prospective, multi-center, single-arm, non-randomized, non-blinded, observational study to evaluate the test-retest reliability of the Visibly Vision Test.

Additionally, observational data will be collected to understand whether the subject performs the set-up process correctly and subject comprehension of the patient labeling will also be evaluated.

DETAILED DESCRIPTION:
Potentially eligible subjects who provide informed consent and are confirmed qualified will be presented a room simulating the home environment with, at minimum, a table; pair of internet-connected devices (if subject has not opted to use their own), as well as some common household items. Subjects will then be directed to visit the website clinical.opternative.com and follow instructions on the website to complete vision testing.

Following completion of the first test session, subjects will undergo a series of critical knowledge task questions administered by site staff to evaluate their understanding of the critical aspects of the proposed patient labeling. Subjects will not receive verbal feedback and the study staff will refrain from any non-verbal responses to the answers provided from the subjects.

At least four hours but not more than 72 hours from the completion of the first test, each subject will be asked to return to the testing room, and complete the Visibly Vision Test again, including repeating the on-boarding, set-up, test, and off-boarding processes.

Site staff will observe and document the second testing process in the same manner as for the subject's first test session.

Following completion of the second test (retest), subject participation will be considered complete.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 22 to 55 years at the time of consent;Recent (within 24 months) in-person comprehensive eye examination with a licensed eyecare professional and have prior prescription values (sphere, cylinder, axis) available;Subject must have either documented recent refractive error not greater than -1.00D of myopia and no greater than -2.00D astigmatism in either eye or documented prior correction no greater than -6.00D of myopia in either eye. Subject are without known existing eye disease or history of systemic disease that may affect the eye; Subjects with known BCVA of 20/32 or better per recent prescription

Exclusion Criteria:

* Subject has had prior use of the Visibly Vision Test; Subjects with known diabetes mellitus; Subjects using ophthalmic or systemic corticosteroids; Subjects with known autoimmune conditions (e.g. Grave's disease, rheumatoid arthritis); Subjects with active corneal or conjunctival infection;Subjects with active corneal, conjunctival, or intraocular inflammation (i.e., uveitis); Subjects with known diabetic retinopathy; Subjects with known glaucoma or ocular hypertension; Subjects with known macular degeneration; Subjects with previous ocular surgery; Subjects using antihyperglycemic agents; corticosteroids; hydroxychloroquine (Plaquenil) and chloroquine (Aralen); tamoxifen (Nolvadex); Subjects with a history of measured spherical difference between left and right eye of 4.00 D or greater;

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Test-retest variability (repeatability) of the Visibly Vision Test in the measurement of refractive error as assessed by the repeatability standard deviation using the Visibly software numerical outputs of estimated refractive error/correction. | Retest conducted between four and 72 hours after initial test.
  The refractive error measurements will be those given by the Visibly software numerical outputs of estimated refractive error/correction.
  For each component of the refractive error measured in diopters (sphere, cylinder, and spherical equivalent), the homogeneous repeatability will be assessed using repeated measurements within study eyes.

SECONDARY OUTCOMES:
Collection of subject comprehension of critical aspects of patient labeling using subject response forms. | Performed immediately after initial test completion
  Collection of response from subjects regarding their comprehension of critical aspects of patient labeling.

CONTACTS AND LOCATIONS:
Locations (1):
- TRA, Harlingen, Texas, United States

IPD SHARING:
Plan to Share IPD: No